CLINICAL TRIAL: NCT00398710
Title: A Phase II Study of Perifosine in Patients With Relapsed/Refractory Waldenström's Macroglobulinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Perifosine 221
Record Dates: First submitted 2006-11-09; First posted 2006-11-14 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2011-11

CONDITIONS: Waldenström's Macroglobulinemia
Keywords: Waldenström's Macroglobulinemia; Perifosine
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — perifosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perifosine (Experimental): Patients will receive perifosine orally at 150 mg daily after food for 28-d cycles.
  Interventions: Drug: Perifosine

INTERVENTIONS:
Drug: Perifosine — 150 mg daily (100 mg daily in case of dose reduction)
  Other Names: D-21266; KRX-0401

SUMMARY:
This is a phase II study in relapsed/refractory WM patients treated with perifosine. It is designed to assess the proportion of overall confirmed responses (CR + PR + MR) using a two-stage phase II study design to permit early stopping of the trial if there is strong evidence that the study regimen is inactive. In addition, it will assess toxicity of this drug in patients with WM. Patients will receive perifosine 150 mg qhs daily. Patients will be assessed by serum immunoelectrophoresis and IgM level at least every 4 weeks.

DETAILED DESCRIPTION:
This is a phase II study in relapsed/refractory WM patients treated with perifosine. It is designed to assess the proportion of overall confirmed responses (CR + PR + MR) using a two-stage phase II study design to permit early stopping of the trial if there is strong evidence that the study regimen is inactive. In addition, it will assess toxicity of this drug in patients with WM. Patients will receive perifosine 150 mg qhs daily. Patients will be assessed by serum immunoelectrophoresis and IgM level at least every 4 weeks.

Patients will take three 50 mg tablets of perifosine qhs daily (for 28 days cycles) with food. Patients may need anti-emetics and/or anti-diarrheas. All patients should continue therapy unless disease progression is documented on two occasions at least 1 week apart. Patients with progressive disease or who refuse further therapy will be discontinued from the protocol. Dose modifications for toxicity will be performed.

Standard criteria for evaluation of response in WM recommended by the Second International WM Workshop will be used in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years.
* Must have received prior therapy for their WM and have relapsed or refractory WM. Any number of prior therapies is acceptable.
* Measurable disease, defined as presence of immunoglobulin M (IgM) paraprotein with a minimum IgM level of > 2 times the upper limit of each institution's normal value is required and over 10% of lymphoplasmacytic cells in the bone marrow.
* ECOG Performance Status (PS) 0, 1, or 2.
* The following laboratory values obtained 14 days prior to registration
* ANC >= 1 x109/L
* PLT >= 75 x109/L
* Total bilirubin ≤ 2.0 mg/dL (If total is elevated check direct and if normal patient is eligible.)
* AST <= 3 x upper limit of normal (ULN)
* Creatinine <= 2 x ULN
* Ability to provide informed consent.
* Life expectancy >= 12 weeks.

Exclusion Criteria:

* Uncontrolled infection.
* Other active malignancies.
* CNS involvement.
* Cytotoxic chemotherapy ≤ 3 weeks, or biologic therapy ≤ 2 weeks, or corticosteroids ≤ 2 weeks, prior to registration. Patients may be receiving chronic corticosteroids if they are being given for disorders other than WM such as auto-immune diseases. Plasmapheresis is not considered as an active therapy and can be used at the physician's discretion.
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational.
* Any of the following:
* Pregnant women
* Nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device (IUD), or abstinence, etc.)
* Known to be HIV positive.
* Radiation therapy ≤ 2 weeks prior to registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-10; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Response rate | Every 4 weeks
  Response will include complete remission, partial remission (PR), and minimal response (MR) using serum protein electrophoresis. Response will also be assessed by IgM using nephelometry.

SECONDARY OUTCOMES:
Safety | Every 4 weeks
  Adverse events will be assessed at each visit and graded according to the National Cancer Institute Common Toxicity Criteria (version 3.0) from the first dose until 30 d after the last dose of perifosine.
Time to progression | Every 4 weeks
  This will be calculated using Kaplan-Meier methodology.
Progression free survival | Every 4 weeks
  This will be calculated using Kaplan-Meier methodology.
Duration of response | Every 4 weeks
  This will be reported among responding patients.

CONTACTS AND LOCATIONS:
Overall Officials: Irene M Ghobrial, MD, Study Chair — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Result] Ghobrial IM, Roccaro A, Hong F, Weller E, Rubin N, Leduc R, Rourke M, Chuma S, Sacco A, Jia X, Azab F, Azab AK, Rodig S, Warren D, Harris B, Varticovski L, Sportelli P, Leleu X, Anderson KC, Richardson PG. Clinical and translational studies of a phase II trial of the novel oral Akt inhibitor perifosine in relapsed or relapsed/refractory Waldenstrom's macroglobulinemia. Clin Cancer Res. 2010 Feb 1;16(3):1033-41. doi: 10.1158/1078-0432.CCR-09-1837. Epub 2010 Jan 26. PMID 20103671